CLINICAL TRIAL: NCT07162727
Title: "Efficacy of Non Perforated Titanium Foil Versus Collagen Membrane on Guided Bone Regeneration for Ridge Augmentation"
Brief Title: Comparison of Non Perforated Titanium Foil Over Collagen Membrane in Ridge Augmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Collaborators: SVS Institute of Dental Sciences (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, Professor and head of the department, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/3/2022
Record Dates: First submitted 2025-08-30; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Ridge Augmentation
Keywords: Alveolar ridge augmentation; Bone height; Bone width; Bone density

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- titanium foil in ridge augmentation (Experimental): Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge defect. HA graft was placed onto the external defect upon which preformed titanium foil (Ti-foil®, India) depending on the size and extent of defect was placed. Foil was stabilized with the help of stainless steel screws of diameter 1.5 cm and length varied depending on the depth of the defect. The flaps were approximated and sutured without tension. Periodontal dressing was given.
  Interventions: Device: titanium foil in ridge augmentation
- collagen membrane in ridge augmentation (Active Comparator): Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge defect. HA graft was placed onto the external defect upon which preformed collagen membrane depending on the size and extent of defect was placed. The flaps were approximated and sutured without tension. Periodontal dressing was given.
  Interventions: Device: collagen membrane

INTERVENTIONS:
Device: titanium foil in ridge augmentation — Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge defect. HA graft was placed onto the external defect upon which preformed titanium foil depending on the size and extent of defect was placed. Foil was stabilized with the help of stainless steel screws of diameter 1.5 cm and length varied depending on the depth of the defect. The flaps were approximated and sutured without tension. Periodontal dressing was given.
  Arms: titanium foil in ridge augmentation
Device: collagen membrane — Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge defect. HA graft was placed onto the external defect upon which preformed collagen membrane depending on the size and extent of defect was placed. The flaps were approximated and sutured without tension. Periodontal dressing was given.
  Arms: collagen membrane in ridge augmentation

SUMMARY:
Aim & Objectives: The aim of the present study was to clinically and radiographically evaluate the efficacy of titanium foil and collagen membrane in ridge augmentation.

Patients and methods: 18 subjects participated in this study. One site in each subjects was randomly assigned into each of the following experimental groups; Test group: ridge augmentation with titanium foil and control group: ridge augmentation with collagen membrane. Radiographic parameters included bone height, bone width and bone density. Evaluations of these parameters were performed after 3 months and 6 months by using Dentium Rainbow software & [reg]. Clinical parameters included the evaluation of Early Healing Score (EHS) during post operative healing period at 1 week and 1 month.

DETAILED DESCRIPTION:
Dental extractions can result in the loss of alveolar bone, leading to a decrease in both bone height and width, which may limit space for implant placement, particularly when taking aesthetic and prosthetic aspects into account.1 Various techniques have been developed for augmenting alveolar ridges, includes Guided Tissue Regeneration (GTR), Guided Bone Regeneration (GBR), onlay grafting, Distraction osteogenesis, which utilizes osteoconductive (scaffold-providing), osteoinductive (stimulating bone-forming cells), and osteogenetic (bone-producing cell-containing) properties.2 GBR membrane plays a vital role as a selective barrier that regulates cellular repopulation at the defect site. It prevents the rapid migration of soft tissue cells such as fibroblasts and epithelial cells, which could otherwise hinder bone regeneration. By excluding these cells, the membrane preserves a protected space that supports the slower infiltration and activity of osteogenic cells responsible for bone formation. Positioned between soft and hard tissues, it ensures a favourable environment for targeted bone regeneration by permitting only bone-forming cells to populate the area.3 GBR membranes are mainly categorized based on their degradation characteristics into non-resorbable (N-RES) and resorbable (RES) varieties. N-RES membranes such as titanium meshes, titanium foil and PTFE membranes offer reliable and enduring results. RES membranes are made from either natural or synthetic polymers, including xenogeneic native collagen, polyglycolide and polylactide polymers.4,5 The collagen membrane is utilized in guided bone regeneration because it can stimulate adhesion, chemotaxis and its own degradation along with that of its progenitor.6 The collagen membrane aids in wound healing by stabilizing clots, maintaining wound stability and hemostasis. It also serves as a scaffold that improves primary wound coverage to attract fibroblasts through its chemotactic properties.7,8 Its main drawbacks are rapid degradation rate and lack of stiffness, which can lead to a collapse of the barrier over the bone defect and diminish the space essential for bone regeneration.9,10 To reduce the risk of bacterial colonization at the graft site, the use of non-permeable occlusive titanium barriers (OTB) has recently been proposed as a promising alternative in reconstructive implant surgeries. These titanium barriers are designed to provide a completely sealed environment that effectively isolates the bone graft from the surrounding soft tissue and oral cavity, thereby minimizing microbial contamination. In addition to their superior biocompatibility and structural rigidity, OTBs offer the advantage of enhanced space maintenance and mechanical stability, which are crucial for successful bone regeneration in complex defects.11 This study aims to evaluate the effectiveness of non perforated titanium foil in comparison to traditional collagen membranes in ridge augmentation procedures, assessing their respective abilities to facilitate predictable and successful bone regeneration.

MATERIALS AND METHODS TRIAL DESIGN The trial was designed as randomized controlled clinical trial, to clinically and radiographically evaluate the efficacy of titanium foil and collagen membrane in ridge augmentation.

PARTICIPANTS AND ELIGIBILITY CRITERIA Subjects for the study were selected from the outpatient section of the Department of Periodontology, Sri Venkata Sai Institute of Dental Sciences, Mahbubnagar, Telangana and were followed up for over six months period after the procedures. Approval from Institutional Ethics Committee (SVSIDS/PERIO/4/2022) was obtained and informed consent was taken from the patients.

SELECTION CRITERIA:

Inclusion criteria:

Systemically healthy male and female patients of age >18 years with atropic areas. Class IV (knife edge form with adequate height but in adequate width of alveolar process) and V (flat ridge form with loss of alveolar process) of Cawood and Howell27 classification were included in the study.

Exclusion criteria:

Medically compromised patients, patients <18 years of age, pregnant women, bruxism patients, heavy smokers, patients who underwent chemotherapy, radiotherapy in the past 12 months were excluded.

RANDOMIZATION AND BLINDING Randomization included computerized generation of the allocation sequence in random permuted blocks (block randomization) and blinding was done by assigning the block sites to study groups according to the specified sequence by a second operator who coded the two sites selected from every patient by the first operator into each of the following group. Test (T): Titanium foil group and Control (C): Collagen group. The blind was not broken until this clinical trial was completely finished. The study was designed as a single blind, randomized controlled clinical to evaluate the efficacy of titanium foil and collagen membrane used in guided bone regeneration.

INTERVENTIONS Presurgical protocol Each patient was prepared for surgery with an initial phase-I therapy which includes scaling and root planing (SRP), occlusal adjustment and oral hygiene instructions. On completion of the initial examination and thorough phase-I therapy, the patients were reassessed after 1 week for their oral hygiene compliance. The patients were recalled for the surgical procedure after 2 weeks.

Surgical Procedure:

Titanium foil:

The surgery was performed under local anaesthesia using 2% lidocaine. Surgical access was attained through a mid-crestal incision followed by an intrasulcular incision at the adjacent teeth. Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge defect. HA graft was placed onto the external defect upon which preformed titanium foil (Ti-foil®, India) depending on the size and extent of defect was placed. Foil was stabilized with the help of stainless steel screws of diameter 1.5 cm and length varied depending on the depth of the defect. The flaps were approximated and sutured without tension. Periodontal dressing was given.

Collagen membrane:

Under local anaesthesia using 2% lidocaine, the surgery was performed. Surgical access was attained through a mid-crestal incision followed by an intrasulcular incision at the adjacent teeth. Full thickness mucoperiosteal flap was elevated, to expose the alveolar ridge. HA graft was placed onto the external defect upon which collagen membrane (Fix Gide®) was placed. The flaps were approximated and sutured without tension. Periodontal dressing was given.

Follow-up and postsurgical care Routine postoperative instructions followed by antibiotics (Amoxicillin 500mg + Clavulanic acid 125 mg twice a day for 5 days and Metronidazole 400mg twice a day for 5 days) and analgesics (Ibuprofen 400 mg thrice a day for 5 days) were prescribed. Patients were recalled 1 week after surgery. Periodontal dressings and sutures were removed. Patients were instructed to gently brush the area with a soft bristled toothbrush. Patients were monitored for 1 week, 3 months and 6months. At each of the recall visits, oral hygiene was assessed. Oral hygiene instructions were reinforced.

Surgical re-entry for titanium foil removal The new bone formed was assessed by measuring bone height (BH), bone width (BW) and bone density (BD) using CBCT after 6months. After assessment, foil removal was done. On the day of foil removal, a full thickness mucoperiosteal flap was raised. The titanium foil was removed slowly as it should not disturb the new bone formed. Stainless steel screw was unscrewed followed by lifting up the foil and thus complete foil was removed. Suturing was done to attain the primary closure.

OUTCOMES Primary outcomes CBCT (Dentium Rainbow software, version 1.0.0.0.) images of maxilla or mandible who are undergoing treatment for ridge augmentation were taken at baseline, 3 months and 6 months. CBCT datasets were acquired by using Dentium Rainbow software®, version (1.0.0.0.) at standard parameters. The raw images were exported into Digital Imaging and Communications in Medicine (DICOM) by using the Dentium Rainbow software. Head position was standardized to ensure that axial sections were parallel to the frankfort plane, and sagittal sections were vertical to the axial plane and parallel to the connection of the anterior nasal spine (ANS) and posterior nasal spine (PNS).

A total of 18 partial edentulous areas seeking CBCT evaluation for ridge augmentation were included. Bone height, bone width and bone density were recorded radiographically using CBCT at baseline, 3 months and 6 months BH was measured from the crest of the alveolar ridge to the superior border of the mandibular canal in the mandible or to the floor of the nasal cavity or maxillary sinus in the maxilla. These measurements were recorded in millimeters (mm) at the center of the edentulous region.

BW was measured in the buccolingual dimension at three standardized levels: 1 mm below the crest (crestal level), mid-height of the alveolar ridge, basal bone (near cortical base). These measurements were done perpendicular to the long axis of the alveolar ridge using the ruler tool in the software.

BD was assessed using CBCT grayscale values (GV) as a surrogate for bone mineral density. Although it is not equivalent to Hounsfield Units (HU), relative GV were used for intra-study comparison. A 1 mm² region of interest (ROI) was selected at each measurement level (crestal, middle, and basal). GV values were recorded and averaged for statistical analysis.

Secondary outcomes:

Postoperatively after 1week and 1month, soft tissue wound healing was assessed by using Early Wound Healing Score (EHS) by Marini et al.,12 The EHS scoring was based on the evaluation of clinical signs of re-epthelialzation, hemostasis and inflammation. The sum of the single scores for these three parameters calculates the EHS, which ranges between 0 to 10 points.

STATISTICAL ANALYSIS:

Data was collected and compiled and entered to excel 2016, statistical analysis was done using Statistical Package for Social Sciences (SPSS) version 21, prepared measures ANOVA test was used to compare the parameters at various intervals, paired t test was used for the pair wise intragroup comparison of parameters, intergroup comparison was done using independent t test. Wilcoxen sign rank test was used for the intragroup comparison of EHS and Mann Whitney U test was used for inter group comparison of EHS values. Confidence intervals were set at 95% and values of p<0.05 were interpreted as statistically significant, p≤0.001 as highly significant, and p≥0.05 as not significant.

DISCUSSION A sufficient amount of alveolar bone is essential for the biomechanical support as well as for aesthetic results.13 However, edentulous regions are usually characterized by alveolar bone loss caused by continuous bone resorption that occurs following tooth loss.14,15,16 Several methods, including distraction osteogenesis, GBR, and onlay block grafts, have been proposed to increase the bone volume for dental implant insertion in cases where there are insufficient alveolar ridges.2,4 The primary cause of the collagen membrane's collapse is its lack of stability and stiffness, which can be achieved by using preformed titanium foil. Boyne was the first to restore significant osseous deformities with titanium membrane.17 In GBR, preformed titanium foil membranes act as barrier which has characteristics of impermeability that prevents soft tissue growing into the grafted area.18,19,20 Its rigidity, biocompatibility and ability to adjust at the recipient site are regarded as major advantage.18 The amount of bone regenerated is proportional to the amount of space beneath the membrane.21 The bone regenerated in membrane protected defects, heals in a sequence of steps that stimulates bone formation after tooth loss. After blood clot formation, bone regeneration is initiated by the formation of woven bone along with new blood vasculature at the periphery of the defect. The woven bone is subsequently replaced by lamellar bone. Bone remodelling occurs with new and secondary osteons.22 The present study clinically and radiographically evaluated the efficacy of titanium foil and collagen membrane used in ridge augmentation. Radiographically, there was significant difference in BH and BW in test group where as, non significant in control group. BD quantified in HU were significant in both the groups.

In the present study, on intra-group comparison, in test group there was significant difference in BW from baseline to 3-months and baseline to 6-months with p value (p=0.010*, p=0.002*) respectively where as 3-months to 6-months there was no significant difference (p=0.052). This was in accordance with the study conducted by Maeda et al.,20 in which they evaluated the combined use of a bovine-derived bone graft and an anodized titanium foil (T Seal) for the reconstruction of compromised alveolar sockets and demonstrated that this combination is highly effective in promoting horizontal bone regeneration. Within six months postoperatively, patients showed significant improvements in the BW and contour of the alveolar crest. The rigid nature of the titanium foil provided excellent space maintenance and protection for the graft material during healing. Additionally, the biocompatibility of both the graft and barrier contributed to favourable tissue responses and predictable outcomes.

In the present study on intragroup comparison, in test group there was significant difference in BH from baseline to 3-months and baseline to 6-months (p=0.003*, p=0.009*) respectively but 3-months to 6-months there was no significant difference (p=0.087) seen. Bassi et al.,23 evaluated the histological and histomorphometric outcomes of preformed titanium foil (PTF) in GBR for posterior mandibular atrophies. Histological analyses demonstrated new bone formation and integration with the graft material, indicating the effectiveness of PTF in vertical bone regeneration.

A study conducted on rabbits by Lundgren et al.,24 concluded that employing a completely occlusive and rigid titanium barrier can effectively facilitate the augmentation of intramembranous bone beyond natural skeletal boundaries. This approach demonstrates the potential for predictable bone regeneration in areas requiring vertical augmentation.

A similar study done in humans and rabbits by Steenberghe et al.,25 demonstrated that occlusive titanium barrier achieved significant bone augmentation. The technique demonstrates the potential for large-volume bone regeneration, providing a viable option for patients with severe bone resorption In the present study, on intragroup comparison BD which is quantified in HU showed highly significant difference in test group (p<0.001**) and significant difference seen in control group (p=0.025*). Milillo et al.,26 used a customized occlusive titanium barrier in GBR, combined with a blood clot and β-TCP filler, proved effective in increasing bone volume to facilitate implant placement. This technique offers a viable alternative to traditional grafting methods, reducing the need for autologous bone harvesting and associated morbidity.

Contrary to the present study, Jung et al.,27 demonstrated the combination of porous titanium mesh with a cross-linked collagen membrane in GBR. Bone density was measured using the Hounsfield scale on cone-beam computed tomography (CBCT) before titanium mesh removal and found that the addition of a collagen membrane improved bone quality and reduced soft tissue interposition over the titanium mesh. In this present study along with collagen membrane, titanium foil also has significant gain in bone density.

In the present study on intergroup comparison, we have observed that BW is non significant at baseline (p=0.27) but there is significant difference seen at 3-months (p=0.049*) and 6-months (p=0.05*). Leiva-Gea et al.,28 evaluated the use of titanium occlusive barriers in guided bone regeneration for horizontal bone augmentation, revealed that this approach yields more reliable and consistent results, with substantial bone volume gains that enhance the success of implant placement.

In the present study on intergroup comparison, BH was analysed and compared between the groups. It showed that there was no significant difference at baseline, 3-months, 6-months (p=0.93, p=0.737, p=0.443). Contrary to the present study, Perret et al.,11 demonstrated that vertical bone augmentation using occlusive titanium barriers is a feasible and effective technique, particularly for severely resorbed alveolar socket and highlighted the advantages of rigid, non-resorbable barriers in providing superior space maintenance and mechanical stability, essential for successful vertical GBR. This method proved especially beneficial in cases where conventional techniques may fail to maintain graft volume or contour. Additionally, the combination with secondary healing was shown to reduce early membrane exposure and support stable tissue regeneration, reinforcing the value of titanium barriers in complex vertical bone augmentation procedures.

In the present study on intergroup comparison, test group reveals that horizontal bone augmentation often yields more predictable outcomes than vertical augmentation in GBR, particularly when utilizing titanium foil. Titanium foil offers excellent mechanical stability, rigidity, space maintenance and formability, making it ideal for contouring over horizontal defects. This allows for the creation of a stable, tented space that resists soft tissue collapse and effectively maintains the graft material in position. In contrast, vertical augmentation poses greater challenges due to gravitational forces, which can displace graft material. limited blood supply at vertical sites, especially in atrophic ridges, soft tissue tension over vertically augmented areas, increasing the risk of wound dehiscence and membrane exposure.63 Similarly in a study done by Perret et al.,29 demonstrated the use of occlusive titanium barriers in GBR for vertical jaw defects and there were predictable and effective outcomes in both hard and soft tissue augmentation. The two-stage approach yielded significantly greater vertical and horizontal bone gains compared to the one-stage approach. Additionally, a spontaneous increase in soft tissue thickness was observed, potentially enhancing long-term implant stability. The study supports the viability of OTBs as a reliable alternative to traditional non-resorbable membranes, offering advantages in cases of accidental exposure and simplifying surgical procedures through pre-shaped designs.

In the present study on intergroup comparison BD which is measured in HU, test group shows significant difference in 3-months and 6-months than baseline, which aligns with the case series done by Bassi et al.,30 where they evaluated the clinical outcomes of using a PTF for GBR in patients with posterior mandibular atrophy and also focused on assessing the effectiveness of PTF in facilitating bone volume augmentation to support dental implant placement The results suggest good potentialities of this method for bone volume augmentation in distal mandibular atrophies, allowing to maximize the outcome and simplifying the surgical phase.

In a similar study by Bassi et al.,19 demonstrated the use of a PTF in GBR for severe mandibular atrophy showing promising results, with substantial bone regeneration and successful implant placement. The technique allowed for precise adaptation to the defect site, maintained space for bone growth, and simplified the surgical procedure. These findings suggest that PTF can be an effective alternative to traditional GBR membranes, especially in complex cases involving significant bone loss.

Gaggl et al.,31 concluded that the use of titanium foil as a barrier membrane in guided bone regeneration (GBR) is an effective method for reconstructing peri-implant bone defects. Their study demonstrated significant vertical and horizontal bone gain, as well as long-term stability of the regenerated bone around dental implants. The rigidity and biocompatibility of titanium foil provide excellent space maintenance and protection of the graft material during healing.

In this study, during second surgery implants were placed simultaneously after titanium foil removal. Out of 9 augmented sites 3 sites were placed with implants. Previous studies on the use of perforated titanium membranes have shown good clinical outcomes, but the presence of perforations exposed the membranes to a greater risk of infection.65 In this study preformed titanium foils act as a total barrier, preventing soft tissue (epithelial and connective tissue) from infiltrating the bone defect, which could otherwise interfere with bone regeneration. This property also makes the titanium foil removal easier during second surgery.

Perret et al.,32 stated that the White Layer Approach offers a simplified, less invasive method for soft tissue augmentation following vertical GBR with OTBs. By utilizing the body's natural healing processes and the formation of pseudo-periosteum, clinicians can achieve significant gains in vertical bone height and soft tissue without additional grafting procedures.

This study presents certain limitations. One of the primary disadvantages of using titanium foil is, it is non-resorbable and needs a second surgical procedure for removal. Another common complication associated with titanium foils is membrane exposure. While the stiffness is beneficial in maintaining space for bone regeneration more effectively than other membranes, it can also lead to mucosal irritation and subsequent exposure. Another issue is the risk of bacterial contamination on exposed titanium surfaces, which may negatively affect wound healing. Therefore, strict oral hygiene protocols are crucial to prevent infection and ensure successful outcomes. To enhance treatment predictability and clinical success, modifications in surgical techniques for alveolar ridge augmentation are needed.32 Additionally, this study reflects short-term clinical outcomes, and the long-term efficacy and biocompatibility of titanium foil should be evaluated in future investigations.

In this study, exposure of the titanium foil occurred in two cases. However, it was observed that both early and late exposures, when managed with proper hygiene, did not compromise the regenerative outcomes. Notably, early exposure contributed to an increase in the thickness of attached gingiva, attributed to secondary intention healing. Finally, it is important to note that no histological analyses were performed in this study, which limits the understanding of the underlying biological processes involved in tissue regeneration.

Within the limitations of the study, we have observed that the use of an PTF can lead to better hard tissue augmentation compared to collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients of age >18 years with atropic areas.
* Class IV (knife edge form with adequate height but in adequate width of alveolar process) and V (flat ridge form with loss of alveolar process) of Cawood and Howell27 classification.

Exclusion Criteria:

* Medically compromised patients
* patients <18 years of age
* pregnant women
* bruxism patients
* heavy smokers
* patients who underwent chemotherapy, radiotherapy in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
bone height | 6 months
  BH was measured from the crest of the alveolar ridge to the superior border of the mandibular canal in the mandible or to the floor of the nasal cavity or maxillary sinus in the maxilla. These measurements were recorded in millimeters (mm) at the center of the edentulous region.
bone width | 6 months
  Bone width was measured in the buccolingual dimension at three standardized levels: 1 mm below the crest (crestal level), mid-height of the alveolar ridge, basal bone (near cortical base). These measurements were done perpendicular to the long axis of the alveolar ridge using the ruler tool in the software.
bone density | 6 months
  Bone density was assessed using CBCT grayscale values (GV) as a surrogate for bone mineral density. Although it is not equivalent to Hounsfield Units (HU), relative GV were used for intra-study comparison. A 1 mm² region of interest (ROI) was selected at each measurement level (crestal, middle, and basal). GV values were recorded and averaged for statistical analysis.

SECONDARY OUTCOMES:
early healing score | 1 month
  Postoperatively after 1week and 1month, soft tissue wound healing was assessed by using Early Wound Healing Score (EHS) by Marini et al.,12 The EHS scoring was based on the evaluation of clinical signs of re-epthelialzation, hemostasis and inflammation. The sum of the single scores for these three parameters calculates the EHS, which ranges between 0 to 10 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Svs Institute of Dental Sciences, Mahbūbnagar, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: IN 2026